CLINICAL TRIAL: NCT06372028
Title: tVNS-combined Motor Training for the Rehabilitation of the Upper Limb in Children and Young People With Cerebral Palsy: a Randomized, Sham-controlled Trial
Brief Title: Non Invasive Vagus Nerve Stimulation in Cerebral Palsy (BOOSTTVNS)
Acronym: (BOOSTTVNS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 944/A
Record Dates: First submitted 2024-04-02; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy
Keywords: transcutaneous Vagus Nerve Stimulation; intensive bimanual training; neurorehabilitation; non invasive brain stimulation; upper limb motor deficit
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tVNS combined with the training (Experimental): The active stimulation will be applied through an active electrode placed on the cymba conchae (the auricular branches of the vagus nerve) of the left ear. The intensity will be set based on the individual perceptual threshold, below the perception of pain. The intensity of the stimulation will be gradually increased in order to reach the intensity of stimulation with a ramping-up phase of 30 secs. The tVNS will be applied for the first 75 minutes of the training, every day of the treatment. Before, 20 minutes and 75 minutes after the start of the stimulation SpO2 and HR will be checked. At the end of the stimulation session participants will be asked to report the sensations and possible side effects occurring during tVNS and to rate their feeling on several visual analogue scales and Likert scales. The intensive bimanual training will be administered by following the procedure described in the Detailed Description session, as for the Sham tVNS combined with the training arm.
  Interventions: Device: transcutaneous vagus nerve stimulation (tVNS)
- Sham tVNS combined with the training (Sham Comparator): The sham stimulation will be applied through an active electrode placed on lobe of the left ear that is free of cutaneous vagal innervations. The stimulation intensity will be set based on the individual perceptual threshold, below the perception of pain. The intensity of the stimulation will be gradually increased in order to reach the intensity of stimulation with a ramping-up phase of 30 secs. The tVNS will be applied for the first 75 minutes of the training, every day of the treatment. Before, 20 minutes and 75 minutes after the start of the stimulation SpO2 and HR will be checked. At the end of the stimulation session participants will be asked to report the sensations and possible side effects occurring during tVNS and to rate their feeling on several visual analogue scales and Likert scales. The intensive bimanual training will be administered by following the procedure described in the Detailed Description session, as for the Active tVNS combined with the training arm.
  Interventions: Device: transcutaneous vagus nerve stimulation (tVNS)

INTERVENTIONS:
Device: transcutaneous vagus nerve stimulation (tVNS) — tVNS allows the non-invasive stimulation of the Vagus Nerve by delivering electrical pulses to the sensory afferent fibers of the auricular, thick-myelinated, branch of the vagus nerve in the outer ear. TVNS seems to engage the same neural pathways of invasive VNS methods and may provide a novel, bottom-up NIBS method to enhance gamma-aminobutyric acid and Noradrenaline levels, which play a pivotal role in brain plasticity. The stimulation will be performed by using a Conformite Europeenne (CE) marked tVNS device tVNS®E (tVNS, technologies Gesellschaft mit beschränkter Haftung (GMBH), Erlangen, Germany). It consists in a programmable stimulation unit connected to two titan ear electrodes that are mounted on a gel frame, allowing to generate and transfer electric impulses from the stimulation unit to the surface of the skin, where the electrodes are applied.

SUMMARY:
The present study aims to assess, through a randomized controlled trial (RCT), the efficacy of transcutaneous Vagus Nerve Stimulation (tVNS) in enhancing the functional changes due to an intensive motor training in children and adolescents with Cerebral Palsy (CP). Particularly, in two different groups active or sham tVNS will be paired with the Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) and we will assess the effects on the upper limbs motor ability and daily functioning in 6 to 17 years old patients with CP having mild-to moderate upper limb deficits. The investigators hypothesized that, thanks to the intensive bimanual training, both the active and the sham group will improve in motor functioning. However, taking into account that tVNS has the potential to facilitate in a bottom-up way neural plasticity, particularly in chronic disease conditions, the investigators hypothesized that active tVNS might improve in a greater and more lasting extent than sham tVNS the motor functioning. Moreover, as suggested by previous studies investigating the effect of non-invasive brain stimulation (NIBS) in paediatric population, the investigators expected that the treatment will be safe and well tolerated. Such a result would encourage the use of NIBS to boost the rehabilitative training of motor abilities in children and adolescents with CP.

DETAILED DESCRIPTION:
This represents one of the two RCTs of the project "Bottom-up and tOp-down neuromOdulation of motor plaSTicity in cerebral palsy" (BOOST; FRRB 3438840). The study will be a randomized, sham controlled, pre-test/post-test study involving 44 children and adolescents with CP. Patients will be treated in pairs, with a matching of motor deficit severity, IQ, and age. Each pair will be randomly assigned to the active or to the sham tVNS group, stratifying the pairs between the two groups based on motor deficit severity, IQ, and age. Both groups will undergo a bimanual training in an ecological and highly motivating environment during the application of the tVNS. During the training, starting from a set of proposals the choice of the type of activities to be practiced in each session will be left to patients, boosting the motivational aspect of the training. This will also ensure an individualized and goal directed approach. The therapists will monitor and modify the activities within each pair to ensure that the intervention maintains the quality of the individualized intervention. The positions performed during bimanual tasks and the activities of daily living will be designed to systematically engage postural control of the trunk and lower limbs according to Habit-ILE protocol. The rehabilitation treatment will be carried out for 5 consecutive days for 3h/day for 2 weeks (30 hours of intervention overall). Children and adolescents will be assessed before the start of treatment (T0), immediately after the end of intensive treatment (T1) and three months after the end (T2). The overall RCT will be structured as follows. In the first session prior the beginning of the training (t0), the RCT will include the administration of all clinical assessment measures and the patients will be asked to perform for 10 minutes an ad-hoc computer based Visuomotor task (please refer to the outcome sessions for more detailed description). Then, patients will undergo the 10 days treatment. For each training day, the treatment will last three hours. During the first 75 minutes of treatment the active or sham tVNS (according to the group allocation) will be delivered. Before starting, 20 minutes after and soon after the end of the stimulation the vital parameters will be checked. After the end of the stimulation, patients will be also asked to rate the sensations experienced during the stimulation through Visual Analogue Scales and through child-friendly Likert scales. Then, they will continue the training for the remaining session time without stimulation. Soon after the end of all the training sessions, patients will carry the t1 evaluation. As for the t0 session, this session will include the administration of the clinical assessment measures and execution for 10 minutes of the Visuomotor task. Three months after the end of the training (t2) the follow up assessment will be conducted, following the same exact procedure of t0.

Primary outcomes will include the following clinical measures: the Assisting Hand Assessment (AHA), the Box and Block Test (BBT) and the performance at the Visuomotor task. Secondary outcomes will include the scores at the following tests: the Children's Hand Experience Questionnaire (CHEQ), the Canadian Occupational Performance Measure (COPM), the Gross Motor Function Measure (GMFM-66); the Melbourne Assessment-2 (MA2) scale, the Vineland Adaptive Behavior Scale Version 2 (VABS II), the Pediatric Quality of Life Inventory (PEDS-QL). Vital parameters (the oxygen saturation (SPO2) and the Heart Rate (HR)), and the scores at the questionnaires assessing stimulation- induced sensations will be also checked to assess the safety and the tolerability of the stimulation. Lastly, the feasibility and the acceptability of the training will be assessed by considering, respectively, the number of patients completing the training/the number of sessions for each patient and the response to ad hoc questionnaires for the patients and their guardians.

All primary and secondary outcomes will be collected at each time point, except for the PEDS-QL and VABS II, which will be administered only at T0 and T2. Furthermore, vital parameters and the questionnaires assessing stimulation-induced sensations will be examined during each stimulation session. The acceptability questionnaires will be administered only after the end of the training (t1).

The patients and their guardians, the personnel responsible for conducting the bimanual training and analysing clinical data will be kept blind to the group allocation. Instead, the coordinator of the study, the staff who will apply the tVNS will be "not blind". With respect to the clinical assessment, whenever possible the staff administering and scoring the scales will be blinded to group allocation. Questionnaire scores and neuropsychological tests will not contain personal information about the subjects, who will be identified by an alphanumeric code. All records that contain names or other personal identifiers, such as informed consent forms, will be stored separately from study records identified by code number. In order to uphold the overall quality of the clinical trial, instances of code breaks should be limited to exceptional circumstances, where knowledge of the actual treatment is deemed absolutely necessary for the ongoing management of the patient.

The intensive treatment will take place at IRCCS E. Medea "Associazione La Nostra Famiglia" in Bosisio Parini (Lecco), at Fondazione Mondino IRCCS (Pavia) and at ASST Ospedali Civili di Brescia.

This trial is supported by Fondazione Regionale per la Ricerca Biomedica (Regione Lombardia), project FRRB 3438840 BOOST "Bottom-up and tOp-down neuromOdulation of motor plaSTicity in cerebral palsy"

ELIGIBILITY:
Inclusion Criteria:

* clinical signs of unilateral or bilateral upper limb deficits (with a difference at least of 25% between more affected and less affected hand at Box and Block test);
* Magnetic Resonance Imaging (MRI) confirmed diagnosis according to Surveillance of Cerebral Palsy (SCPE) criteria;
* Manual Ability Classification System (MACS) level I,II,III;
* Gross Motor Function Classification System (GMFCS) level I,II,III;
* Visual Function Classification System (VFCS) I-II-III;
* Intelligence quotient (IQ) > 50.

Exclusion Criteria:

* presence of cochlear implant, cardiac pacemaker, ventriculoperitoneal shunt, neuro-stimulators, clips, fragments or metal splinters in the brain or skull except for titanium;
* treatments for spasticity or functional surgery of the upper limb in the previous 6 months or planned during the duration of the study;
* uncontrolled epileptic seizure in the last 2 years.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Assisting Hand Assessment (AHA) | 1-2 days before the start of training (t0), 1-2 days after the end of the training (t1), three months after the end of the training (t2)
  This scale enables to quantify the assistance provided by the more affected hand to the less affected hand during bimanual activities. This observation-based, criterion-referenced assessment highlights a person's typical performance, emphasizing practical functionality over maximal capacity, and serves as a reliable measure of change over time. The scale comprised 20 items, scored on a 4-point Likert scale, from 1 to 4. The total score indicates how well the more affected hand is used as an assisting hand. A score of 20 means poor performance (the hand is not used as an assisting hand); a score of 80 means that the hand is used effectively. The results are converted for each of the three scales to logits by a Rasch analysis, on a 0-to-100 scale (with higher scores suggesting better use).
Box and Block Test (BBT) | 1-2 days before the start of training (t0), 1-2 days after the end of the training (t1), three months after the end of the training (t2)
  This test is designed to measure manual dexterity. It is quick, simple, and cost-effective. It involves a box with a partition in the middle placed on a table, with a total of 150 blocks on one side of the partition. The score of the test is given by the number of blocks transported within a minute. Higher values suggest better performance. The BBT provides a reliable and objective measurement of manual dexterity, making it valuable for evaluating functional outcomes and monitoring progress in rehabilitation programs over a short period of time.
Visuomotor task | 1-2 days before the start of training (t0), 1-2 days after the end of the training (t1), three months after the end of the training (t2)
  The visuomotor task is an ad hoc computer based task. It involves a mouse click-and-drag operation where an object appears at the center of the screen. The objective is to drag and drop the object to the location indicated by a previously presented arrow, pointing towards a target object within a configuration of objects. Participants are required to focus on the arrow's direction, swiftly and accurately moving the central object to its designated target location. This task enables the measurement of movement time (in milliseconds; consisting in the time necessary to move the object in the target position); precision error (calculated as the distance, in pixels, between the drop position of the object and the actual target position); the proportion of overtime errors (the percentage of trials in which responses are too slow). Smaller values of Movement time, Precision error and overtime errors will suggest better performance.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 1-2 days before the start of training (t0), 1-2 days after the end of the training (t1), three months after the end of the training (t2)
  This is a client-centered, semi-structured interview used in occupational therapy to identify the problems experienced by the patients. This interview engages the patient in recognizing daily occupations of importance that he/she want to do, need to do, or are expected to do but is unable to accomplish. Upon the identification of the problems experienced in patient's everyday-life activities, the patient is asked to rate the importance of each activity in his/her life though a 10-point rating scale and then, to select up to five problems to be addressed during the intervention. Lastly, the patient is asked to rate on a 10-point scale his/her own level of performance and satisfaction in performing that activity for each of the five problems (from 0, low performance or low satisfaction to 10, high performance or high satisfaction).
Children's Hand-UseExperienceQuestionnaire (CHEQ) | 1-2 days before the start of training (t0), 1-2 days after the end of the training (t1), three months after the end of the training (t2)
  The questionnaire includes 27 bimanual activities. Each activity is rated on three scales measuring: i) the perceived efficacy of the activity ("How do you think the child's hand works?") from 1 (Bad / not used hand) to 4 (Good efficacy); ii) the amount of assistance and the time needed to perform the activity ("How much time does your child need to do the whole task, compared to peers?) from 1 (Considerably longer) to 4 (Equally long time compared to other peers); and iii) the child's satisfaction with their performance ("Is your child bothered by his/her reduced hand/arm function during this activity?") from 1 ("It bothers him/her a lot") to 4 ( "It does not bother him/her at all"). The questionnaire provides a result corresponding to the summary of the ratings. The results are converted for each of the three scales to logits by a Rasch analysis, on a 0-to-100 scale (with higher scores suggesting better performance/satisfaction).
Melbourne Assessment 2 (MA2) | 1-2 days before the start of training (t0), 1-2 days after the end of the training (t1), three months after the end of the training (t2)
  This scale allows evaluating the unimanual performance of both the more and less affected hand. It measures four elements of upper limb movement quality: movement range, accuracy, dexterity and fluency. It consists of 14 test items that require children to interact (by reaching, grasping, releasing and manipulating) with simple objects. Movement elements are scored on a 3-, 4-, or -5 point scale according to specific criteria. Scores are arranged into the 4 sub-scales (movement range, accuracy, dexterity and fluency) according to the element of movement being rated. A child's total raw score for each sub-scale is converted to a percentage of the maximum possible score for that sub-scale, with higher scores indicating better performance.
Gross Motor Function Measure (GMFM-66) | 1-2 days before the start of training (t0), 1-2 days after the end of the training (t1), three months after the end of the training (t2)
  It is a standardized observational tool used by healthcare professionals to evaluate and quantify the gross motor abilities and limitations of children with CP. It assesses 66 motor skills across five dimensions: lying and rolling, sitting, crawling and kneeling, standing, and walking, running, and jumping. Each skill is scored on a 4-point scale, ranging from 0 (does not initiate) to 3 (performs fully).
Vineland Adaptive Behavior Scale Version 2 (VABS II) | 1-2 days before the start of training (t0), three months after the end of the training (t2)
  This is a tool designed to assess adaptive behavior in individuals from birth to age 90. It assesses 11 subdomains of adaptive behavior grouped into four domains; sums of these scores are standardized into Communication, Daily Living Skills, Socialization and Motor Skills domain standard scores. Sums of the domain standard scores are then standardized into the Adaptive Behavior Composite score ranging from 20 to 160 (mean=100; standard deviation= 15).
Pediatric quality of life inventory PedsQL(cerebral palsy module), (PEDS-QL) | 1-2 days before the start of training (t0), three months after the end of the training (t2)
  This is a widely employed, brief, and standardized self-reporting tool for assessing health-related quality of life in children and young individuals. The measure can be completed by parents (the Proxy Report) as well as children and young people (the Self-Report) with versions available for children and young people aged 5-7, 8-12, and 13-18. Parent-rated versions are available for children aged 2-4, 5-7, 8-12, and 13-18. The versions from 5 to 18 years comprise 35 items comprising 7 dimensions: Daily Activities; School Activities; Movement and Balance; Pain and Hurt; Fatigue;Eating Activities; Speech and Communication. For each item, consisting in everyday life action, it is required to indicate how much of a problem each item has been in the past month with response options from 0 (never a problem) to 4 (almost always a problem). The items are reverse scored and transformed to a 0-100 scale, with higher scores indicating better health related quality of life.

OTHER OUTCOMES:
Heart rate (HR). | in the first 2 minutes, after 20 minutes of stimulation, after 75 minutes of stimulation
  To assess the safety of the stimulation, the HR (beats per minute, bpm) will be checked. HR values will be check during a two minutes rest condition. For this measure, more caution will be held with values lower than 70 or higher than 120 bpm in 6 to 12 years old children and lower than 60 or higher than 100 bpm in 12 to 18 years old adolescents.
Oxygen saturation (SPO2). | in the first 2 minutes, after 20 minutes of stimulation, after 75 minutes of stimulation
  To assess the safety of the stimulation, the SPO2 (%) will be checked, too. SP02 values will be check during a two minutes rest condition. Cases with SPO2 values lower than 93% will be carefully checked.
Tolerability of the stimulation | immediately after every stimulation sessions of the 10-days training
  Tolerability will be assessed through a 10 centimetres Visual Analogue Scale by asking to indicate the level of discomfort experienced during the stimulation, and to rate on Child-friendly Likert scales the intensity of the following sensations: itching, pain, burning, heat, pinching, iron taste, and fatigue, others. For each sensation the patients will be asked to express a value of perception strength that ranges from 0 (absence) to 4 (strong). Higher values will suggest stronger discomfort.
Number of patients who accept to complete the 2-week training | 1-2 days after the end of the training (t1)
  This value will be expressed as percentage, with respect to the total number of recruited patients. Higher values will suggest higher feasibility of the training.
Number of sessions completed per patient | 1-2 days after the end of the training (t1)
  This value will be expressed as mean percentage of session completed (across patients), with respect to the total number of session planned for the training. Higher values will suggest higher feasibility of the training.
Acceptability of the training | 1-2 days after the end of the training (t1)
  The acceptability will be assessed by asking to the child/adolescent and his/her parents subjective evaluation of training accessibility and efficacy. Questions like "I find it difficult to motivate my child for doing the training"/ "I find it difficult to start the training"; or "I would suggest this training to other people I know"/ "I think other people I know would enjoy doing this training" will be rated from 1 (completely disagree) to 5 (completely agree). Response will be reversed in the negative items, so that higher scores will suggest more positive evaluation/higher acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute, IRCCS E. Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymized dataset will be available at https://osf.io/
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Before data analyses, for ten years.
Access Criteria: all
URL: https://osf.io/

REFERENCES:
- [Derived] Vacchini V, Brafa B, Nicotra R, Capelli E, Signorini S, Gasparroni V, Michelutti A, Oldrati V, Galli J, Urgesi C, Cattaneo Z, Fazzi EM, Borgatti R, Finisguerra A, Orcesi S; Boost Working Group. Improving neuroplasticity and Quality of Life in children with Cerebral Palsy: a customized intensive motor training protocol integrating the HABIT-ILE approach. Front Rehabil Sci. 2025 Oct 13;6:1613103. doi: 10.3389/fresc.2025.1613103. eCollection 2025. PMID 41158535
- [Derived] Oldrati V, Gasparroni V, Michelutti A, Ciricugno A, Borgatti R, Orcesi S, Fazzi E, Morandi A, Galli J, Piccinini L, Maghini C, Arioli M, Cattaneo Z, Urgesi C, Finisguerra A. Pairing transcutaneous vagus nerve stimulation with an intensive bimanual training in children and adolescents with cerebral palsy: study protocol of a randomized sham-controlled trial. Front Neurol. 2024 Aug 16;15:1441128. doi: 10.3389/fneur.2024.1441128. eCollection 2024. PMID 39220734